CLINICAL TRIAL: NCT06298448
Title: Impact of Mepolizumab Treatment on the Nasal Microbiome and Local and Systemic Immune Response in Eosinophilic Granulomatosis With Polyangitis (eGPA)
Brief Title: eGPA and Local Inflammation Within the Ear, Nose and Throat Area
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: NL83176.042.23
Record Dates: First submitted 2024-02-05; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: EGPA - Eosinophilic Granulomatosis With Polyangiitis
MeSH Terms: conditions — Churg-Strauss Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, nasal fluid, stool, urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- eGPA: Eosinophilic granulomatosis with polyangiitis patients before and after treatment with mepolizumab will be compared
  Interventions: Diagnostic Test: laboratory experiments before and after mepolizumab treatment
- GPA: Comparator group not treated with mepolizumab
  Interventions: Diagnostic Test: laboratory experiments before and after mepolizumab treatment
- Asthma: Asthma patients before and after treatment with mepolizumab
  Interventions: Diagnostic Test: laboratory experiments before and after mepolizumab treatment
- CRSwNP: Chronic rhinosinusitis patients before and after treatment with mepolizumab
  Interventions: Diagnostic Test: laboratory experiments before and after mepolizumab treatment
- Healthy: Healthy comparator group
  Interventions: Diagnostic Test: laboratory experiments before and after mepolizumab treatment

INTERVENTIONS:
Diagnostic Test: laboratory experiments before and after mepolizumab treatment — Patients that start with mepolizumab treatment on the basis of the clinical disease course will be measured prior and after start of mepolizumab to evaluate the effects this medication has on various immunological parameters and microbiome

SUMMARY:
Rationale: Eosinophilic Granulomatosis with Polyangiitis (eGPA), eosinophilic asthma and chronic rhinosinusitis with nasal polyps (CRSwNP) are airway diseases where eosinophils and interleukine-5 are involved in the pathogenesis. eGPA differs from the other diseases with respect to involvement of other organs. The investigators hypothesize that nasal microbiome dysbiosis with a central augmenting role for S. Aureus plays an important role in disease expression. The investigators expect that anti-interleukin-5 treatment with mepolizumab restores the changes of the nasal microbiome and immune responses to a healthy control phenotype. To study this, the nasal microbiome, the local and systemic immune response and the effect of mepolizumab treatment will be assessed.

DETAILED DESCRIPTION:
See Brief summary.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age

  * able to give informed consent
  * In CRSwNP group: availability of bilateral nasal polyps as diagnosed by endoscopy or CT scan
  * In Severe asthma group: clinical diagnosis of asthma with forced expiratory volume at one second(FEV1) <80% AND either FEV1 reversibility >12% initial or documented positive metacholine challenge (PC20 < 8 mg/ml)
  * In eGPA group: Fulfilling the 2022 ACR/EULAR criteria for eGPA (Wechsler et al., 2017)
  * In GPA group: fulfilling the American College of Rheumatology (ACR)/EULAR GPA criteria (Robson et al., 2022)
  * In healthy controls: absence of asthma symptoms, no bronchial hyperresponsiveness

Exclusion Criteria:

* unable to give informed consent
* Active smoking < (less than) 6 months from baseline visit
* Concomitant use of dupilumab within 6 months of baseline visit
* pregnant or breastfeeding woman
* in CRSwNP group: current use of asthma medication, eGPA
* in healthy controls: chronic use of local anti-inflammatory agents
* in healthy controls: use of immunosuppressive medication
* in healthy controls: use of antibiotics within the last month (before start study/screening/)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with eosinophil driven inflammation for which mepolizumab might be considered for treatment
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The effect mepolizumab treatment has on the nasal microbiome profiles | three months
  Paired change in microbiome diversity index for patients treated with mepolizumab.

OTHER OUTCOMES:
Exploratory evaluation of between group differences | Through study completion, an average of two years
  Microbiome and immunological gene expression values will be measured and differential expression analysis will be performed
Mepolizumab effect on outcome 2 | Through study completion, an average of two years
  The effect mepolizumab treatment has on the immunological gene expression will be measured by differential gene expression analysis.
s there a correlation between the disease activity, the quality of life and the microbiome and immune parameters? | Through study completion, an average of two years
  Spearman ranks correlation

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Fully anonymized data will be made available for other researchers